CLINICAL TRIAL: NCT00921336
Title: Open-Label, Sequential, Ascending, Multi-Dose, Phase 1 Study of KW-2450 as Monotherapy in Subjects With Previously Treated Advanced Solid Tumor
Brief Title: Safety Study to Evaluate KW-2450 in Subjects With Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2450-US-001
Record Dates: First submitted 2009-05-27; First posted 2009-06-16 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Solid Tumor
Keywords: subjects with advanced Solid tumor who have not responded to standard therapy or for whom no standard therapy is available
MeSH Terms: interventions — KW-2450

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KW-2450 (Experimental)
  Interventions: Drug: KW-2450

INTERVENTIONS:
Drug: KW-2450 — Dose escalation may proceed once >= 3 subjects have completed the Day 29 blood sample to evaluate glucose. The safety of each dose level will be established prior to enrollment of subjects in the next dose level. Dose escalation will proceed sequentially with accelerated escalation. Once the criteria for completing the accelerated titration are reached, dose escalation will follow a modified Fibonacci schedule. Up to 6 subjects will be enrolled at each dose level. Enrollment will proceed until the maximum tolerated dose (MTD) has been established or the highest dose level (800 mg/day) has been reached. The Sponsor will enroll up to 12 additional subjects, in an expanded safety cohort.

SUMMARY:
This study will determine the maximum dose of KW-2450 that can be administered safely to subjects with advanced previously treated solid tumor and evaluate its effectiveness.

DETAILED DESCRIPTION:
This open-label, sequential, ascending, multi-dose, Phase 1 study will enroll up to 72 subjects with previously treated advanced solid tumor. Subjects at each dose level will receive KW-2450 orally, once daily for 28 days followed by a 1-week observation period. After completing the 1 week observation period, all subjects will receive KW-2450 on a continuous daily schedule. All doses of KW-2450 will be administered to subjects under overnight fasting conditions.

Dose escalation may proceed once >= 3 subjects have completed the Day 29 blood sample to evaluate glucose. The safety of each dose level will be established prior to enrollment of subjects in the next dose level. Dose escalation will proceed sequentially with accelerated titration. Once the criteria for completing the accelerated titration are reached, dose escalation will follow a modified Fibonacci schedule. Up to 6 subjects will be enrolled at each dose level. Enrollment will proceed until the maximum tolerated dose (MTD) has been established or the highest dose level (800 mg/day) has been reached.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signed and dated Institutional Review Board (IRB) approved informed consent form and Health Insurance Portability and Accountability Act (HIPAA) authorization in accordance with regulatory and institutional guidelines. This must be obtained before performing protocol-related procedures that are not part of standard subject care
2. Histopathologically- or cytologically-documented, advanced primary or recurrent solid tumor that has not responded to an adequate course of available therapy, that has progressed or recurred despite an adequate course of available therapy, that is not curable by available therapy or for which no accepted standard therapy exists
3. Ability to comply with visits/procedures required by the protocol. Subjects enrolled in this trial must be treated at a participating center
4. A life expectancy of >3 months
5. Eastern Cooperative Oncology Group (ECOG) performance status score of <= 2 at study entry
6. Adequate hematologic function, as defined by:

   an absolute neutrophil count (ANC) >= 1500/mm3 a hemoglobin level >=8.5 gm/dL a platelet count >=100,000/mm3
7. Adequate hepatic function, as defined by:

   a total bilirubin level <= 1.5 x the upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine transaminase (ALT) levels <= 2.5 x the ULN or <= 5 x the ULN if known liver metastases
8. Adequate renal function, as defined by:

   a serum creatinine (Scr) <= 1.5 mg/dL for male subjects; Scr <= 1.40 mg/dL for female subjects Calculated creatine clearance > 60 mL/min based on Cockcroft-Gault formula
9. Subjects must be recovered from the effects of any prior anti-neoplastic therapy. The ongoing adverse events due to these therapies must be <=Grade 1 prior to entering the study. At least 5 half-lives should have elapsed for any investigational agents prior to the administration of study medication
10. Subjects with central nervous system (CNS) metastases are eligible for enrollment if they have received prior radiotherapy and/or surgery to site(s) of CNS metastatic disease, have been off glucocorticoids for at least 4 weeks, are not taking anticonvulsants, and have no overt evidence of neurological deficit
11. Men and women, >= 18 years of age at the time of enrollment
12. Women of childbearing potential (WOCBP) must agree to use effective contraception, defined as oral contraceptives, double barrier method (condom plus spermicide or diaphragm) or abstain from sexual intercourse during the study and for 90 days following the last dose of KW-2450.

    WOCBP include females who have experienced menarche and who have not undergone successful sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal (defined as amenorrhea >= 12 consecutive months)
13. Male subjects must be willing to use an appropriate method of contraception (e.g., condoms) or abstain from sexual intercourse and inform any sexual partners that they must also use a reliable method of contraception (e.g., birth control pills) during the study and for 90 days following the last dose of KW-2450
14. WOCBP must have a negative pregnancy test within 7 days of receiving study medication.

Exclusion Criteria:

1. Women who are pregnant or lactating
2. Known diabetes defined as:

   * random serum glucose concentration of > 200 mg/dL
   * fasting plasma glucose (FPG) of > 126 mg/dL
   * 2-hour post load serum glucose concentration of > 200 mg/dL following an oral glucose tolerance test
   * the need for an oral hypoglycemic agent or insulin in order to keep the serum glucose below the above levels; or
   * any diabetic complication (cataract, retinopathy, nephropathy, etc.).
3. Subjects showing clinical evidence or with a history of cataract(s) or retinopathy
4. Abnormal free T4 values. Abnormal thyroid stimulating hormone (TSH) values at enrollment will be further evaluated by free T4. Subjects with abnormal free T4 values and a history or evidence of thyroid disease will be excluded.
5. Subjects who are unable or unwilling to take metformin
6. Uncontrolled intercurrent illness including, but not limited to:

   * Ongoing or active infection requiring parenteral antibiotics;
   * A serious or nonhealing active wound, ulcer, or bone fracture;
   * Uncontrolled hypertension (systolic blood pressure >160 mm Hg, diastolic blood pressure >100 mm Hg, found on two consecutive measurements separated by a 1week period despite treatment with two antihypertensive agents)
7. Unstable cardiovascular disease (i.e., including uncontrolled ischemic heart disease, congestive heart failure, arrhythmia or hypertension; New York Heart Association >= class III; or myocardial infarction or acute coronary syndrome within 6 months)
8. Positive for human immunodeficiency virus, hepatitis B or C
9. Subjects with inflammatory diseases of the gastrointestinal tract or malabsorption syndrome
10. Major surgery within 4 weeks prior to the administration of study medication
11. Evidence of organ dysfunction or any clinically significant deviation in physical examination, vital signs, or clinical laboratory determination;
12. Prolonged QT intervals or any clinically significant abnormalities on ECG
13. A history of prior treatment with other agents specifically targeting IGFRs
14. Subjects who require pharmacological doses of glucocorticoids beyond replacement doses. The use of topical, intra-ocular or inhalation glucocorticoids is permitted
15. Strong inhibitors/inducers of CYP3A4/5, herbal medications (within 1 week of administration of study medication), or drugs for prevention of graft versus host disease or transplant rejection (within 2 months prior to the administration of study medication)
16. Hematopoetic growth factors and erythropoiesis-stimulating agents within 3 weeks prior to the administration of study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To establish the safety, tolerability, and recommended Phase 2 dose of KW 2450 administered orally in subjects with advanced solid tumor who have not responded to standard therapy or for whom no standard therapy is available | 28 days

SECONDARY OUTCOMES:
To determine the PK/PD profile of KW-2450 | PK/PD perfomed up to Day 29 Tumor assessments performed at 8 weeks
To evaluate for preliminary evidence of efficacy | PK/PD perfomed up to Day 29 Tumor assessments performed at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kurman, MD, Study Director — Kyowa Hakko Kirin Pharma, Inc.
Locations (3):
- United States (3):
  - University of Maryland Greenbaum Cancer Center, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering, New York, New York